CLINICAL TRIAL: NCT01181674
Title: Remission Evaluation of Metabolic Interventions in Type 2 Diabetes (REMIT): A Randomized Controlled Pilot Trial
Brief Title: Remission Evaluation of Metabolic Interventions in Type 2 Diabetes (REMIT Pilot Trial)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Dr. Hertzel Gerstein, Director, Division of Endocrinology and Metabolism, McMaster University, Population Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REMIT Pilot; Control # 139433, 143584 (Other: Health Canada); 10-346 (Other: Hamilton Health Sciences Research Ethics Board)
Record Dates: First submitted 2010-08-11; First posted 2010-08-13 (Estimated); Results first posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes; Insulin; Glargine; Metformin; Acarbose; Diet; Exercise; Lifestyle
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance; Motor Activity | interventions — Insulin Glargine; Metformin; Acarbose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (short) (Experimental)
  Interventions: Drug: insulin glargine; Drug: metformin; Drug: acarbose; Behavioral: lifestyle therapy
- Group 2 (long) (Experimental)
  Interventions: Drug: insulin glargine; Drug: metformin; Drug: acarbose; Behavioral: lifestyle therapy
- Standard care (Other)
  Interventions: Other: Standard glycemic care

INTERVENTIONS:
Drug: insulin glargine — sc injection
  Arms: Group 1 (short)
Drug: metformin — oral administration
  Arms: Group 1 (short)
Drug: acarbose — oral administration
  Arms: Group 1 (short)
Behavioral: lifestyle therapy — diet and exercise
  Arms: Group 1 (short)
Drug: insulin glargine — sc injection
  Arms: Group 2 (long)
Drug: metformin — oral administration
  Arms: Group 2 (long)
Drug: acarbose — oral administration
  Arms: Group 2 (long)
Behavioral: lifestyle therapy — diet and exercise
  Arms: Group 2 (long)
Other: Standard glycemic care — as informed by the current clinical practice guidelines
  Arms: Standard care

SUMMARY:
The purpose of this pilot trial is to determine whether an intensive treatment with insulin glargine, metformin, acarbose and lifestyle can normalize blood glucose levels in patients with recently diagnosed type 2 diabetes mellitus when compared to standard diabetes care.

DETAILED DESCRIPTION:
This is a pilot trial of 125 patients allocated to either usual care (1/3), 2 months or 4 months of intensive lifestyle and pharmacotherapy followed by cessation of all drug therapy.

ELIGIBILITY:
Inclusion Criteria:

1. men and women 30-80 years of age inclusive
2. type 2 diabetes mellitus diagnosed by a physician within 3 years prior to patient enrollment
3. anti-diabetic drug regimen (either drug or dose of drug) unchanged during 8 weeks prior to screening and randomization
4. HbA1C ≤ 8.5% on no oral hypoglycemic agents or HbA1C ≤ 7.5% on 1 agent or on half-maximal doses of 2 agents
5. body mass index ≥ 23 kg/m2
6. a negative pregnancy test and an agreement to use a reliable method of birth control for the duration of the trial in all females with childbearing potential
7. ability and willingness to perform self-monitoring of capillary blood glucose (SMBG)
8. ability and willingness to self-inject insulin
9. provision of informed consent.

Exclusion Criteria:

1. current use of insulin therapy
2. history of hypoglycemia unawareness, or severe hypoglycemia requiring assistance
3. renal dysfunction as evidenced by serum creatinine (Cr) ≥ 124 μmol/l
4. history of lactic acidosis or diabetic ketoacidosis
5. active liver disease or elevated alanine transferase (ALT) levels ≥ 2.5 times upper limit of normal at the time of enrollment
6. history of inflammatory bowel disease, colonic ulcers, recent or significant bowel surgery, or predisposition to bowel obstruction
7. cardiovascular disease including any of:

   * systolic blood pressure >180 mmHg or diastolic blood pressure >105 mmHg
   * peripheral vascular disease
   * left bundle branch block or third degree AV block
   * tachyarrhythmias or bradyarrhythmias with uncontrolled ventricular rate
   * stenotic valvular heart disease
   * cardiomyopathy
   * history of heart failure
   * history of aortic dissection
   * documented history of angina or coronary artery disease
   * history of stroke or transient ischemic attack
8. pulmonary disease with dependence on oxygen
9. history of any disease requiring intermittent or continuous systemic glucocorticoid treatment
10. history of any major illness with a life expectancy of <3 years
11. history of injury or any other condition that significantly limits participant's ability to achieve moderate levels of physical activity
12. any history of excessive alcohol intake, acute or chronic
13. known hypersensitivity to metformin, acarbose, or insulin glargine.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2011-01; Primary Completion 2015-02 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hertzel Gerstein, MD, Principal Investigator — Population Health Research Institute; Natalia McInnes (nee Yakubovich), MD, Principal Investigator — Population Health Research Institute
Locations (1):
- McMaster University Medical Centre, Diabetes Care and Research Program, Hamilton, Ontario, Canada

REFERENCES:
- [Result] McInnes N, Smith A, Otto R, Vandermey J, Punthakee Z, Sherifali D, Balasubramanian K, Hall S, Gerstein HC. Piloting a Remission Strategy in Type 2 Diabetes: Results of a Randomized Controlled Trial. J Clin Endocrinol Metab. 2017 May 1;102(5):1596-1605. doi: 10.1210/jc.2016-3373. PMID 28324049

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 (Short) | Group 2 (Long) | Standard Care
Started | 28 | 27 | 28
Completed | 28 | 27 | 26 (28 included in analyses)
Not Completed | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (Short) | Group 2 (Long) | Standard Care | Total
Number analyzed (Participants) | 28 | 27 | 28 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (9.2) | 57.9 (10.5) | 58.2 (11.1) | 57.1 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 14 | 43
  Male | 14 | 12 | 14 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 25 | 23 | 25 | 73
  Non-Caucasian | 3 | 4 | 3 | 10
Region of Enrollment [Number; unit: participants]
  Canada | 28 | 27 | 28 | 83

OUTCOME MEASURES:

1. Primary Outcome: Normoglycemia on Therapy
Description: 1. Percentage of participants achieving normoglycemia on therapy in the experimental group 1 compared to the control group.
  2. Percentage of participants achieving normoglycemia on therapy in the experimental group 2 compared to the control group.
  Normoglycemia on therapy is defined as a mean fasting capillary blood glucose </=5.4 mmol/L and a mean 2-hour pc blood glucose </=6.8 mmol/L on 2 seven-point glucose profiles.
Time Frame: (1) 8 weeks and (2) 16 weeks
Population: Primary outcome (1) is reported in Experimental Group 1 and Standard care at 8 weeks. Primary outcome (2) is reported in experimental Group 2 and Standard care at 16 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Short) | Group 2 (Long) | Standard Care
Number analyzed (Participants) | 28 | 27 | 28
Participants
  Group 1 and Standard care at 8 weeks: number analyzed (Participants) | 28 | 0 | 28
  Group 1 and Standard care at 8 weeks | 14 |  | 1
  Group 2 and Standard care at 16 weeks: number analyzed (Participants) | 0 | 27 | 28
  Group 2 and Standard care at 16 weeks |  | 19 | 1

2. Secondary Outcome: 1) Percentage of Participants With Normal Glucose Tolerance in the Experimental Group 1 Compared to the Control Group. 2) Percentage of Participants With Normal Glucose Tolerance in the Experimental Group 2 Compared to the Control Group.
Description: Normal glucose tolerance is defined as a fasting plasma glucose <6.1 mmol/L and a 2-hour pc plasma glucose <7.8 mmol/L on a 75 g oral glucose tolerance test off diabetes drugs.
Time Frame: (1) 20 weeks and (2) 28 weeks
Population: Outcome (1) is reported in Experimental Group 1 and Standard care at 20 weeks. Outcome (2) is reported in experimental Group 2 and Standard care at 28 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Short) | Group 2 (Long) | Standard Care
Number analyzed (Participants) | 28 | 27 | 28
Participants
  Group 1 and Standard care at 20 weeks: number analyzed (Participants) | 28 | 0 | 28
  Group 1 and Standard care at 20 weeks | 2 |  | 2
  Group 2 and Standard care at 28 weeks: number analyzed (Participants) | 0 | 27 | 28
  Group 2 and Standard care at 28 weeks |  | 2 | 1

3. Secondary Outcome: Percentage of Participants With Normal Fasting Plasma Glucose
Description: Normal fasting plasma glucose is defined as <6.1 mmol/L.
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Short) | Group 2 (Long) | Standard Care
Number analyzed (Participants) | 23 | 23 | 25
Participants | 5 | 5 | 3

4. Secondary Outcome: Change in Fasting Plasma Glucose From Baseline
Time Frame: Baseline and 52 weeks
Population: FPG was not available for some participants at 52 weeks.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Group 1 (Short) | Group 2 (Long) | Standard Care
Number analyzed (Participants) | 23 | 23 | 25
mmol/L | -0.23 (0.96) | -0.64 (1.38) | 0.05 (1.02)

5. Secondary Outcome: HbA1C
Time Frame: 8, 20, 28 and 52 weeks
Population: Some participants did not provide HbA1C values.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Group 1 (Short) | Group 2 (Long) | Standard Care
Number analyzed (Participants) | 24 | 23 | 25
percent
  8 weeks | 6.1 (0.5) | 6.0 (0.4) | 6.6 (0.7)
  20 weeks | 6.2 (0.4) | 6.1 (0.3) | 6.6 (0.7)
  28 weeks | 6.5 (0.8) | 6.4 (0.5) | 6.6 (0.7)
  52 weeks | 6.4 (0.8) | 6.7 (0.7) | 6.5 (0.7)

6. Secondary Outcome: Change in Weight From Baseline
Time Frame: Baseline, 8, 20, 28 and 52 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Group 1 (Short) | Group 2 (Long) | Standard Care
Number analyzed (Participants) | 23 | 22 | 25
kg
  Baseline | 99.5 (23.3) | 95.3 (15.2) | 89.3 (14.6)
  8 weeks | 95.3 (21.8) | 92.4 (15.0) | 87.1 (14.1)
  20 weeks | 92.8 (21.1) | 90.5 (14.8) | 86.3 (13.5)
  28 weeks | 93.3 (20.6) | 91.7 (15.2) | 86.1 (13.5)
  52 weeks | 96.6 (21.7) | 93.8 (16.4) | 86.5 (14.6)

7. Secondary Outcome: Number of Participants With Symptomatic Hypoglycemic Episodes
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Short) | Group 2 (Long) | Standard Care
Number analyzed (Participants) | 28 | 27 | 28
Participants | 9 | 10 | 1

8. Secondary Outcome: Number of Participants With Severe Hypoglycemic Episodes
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Short) | Group 2 (Long) | Standard Care
Number analyzed (Participants) | 28 | 27 | 28
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | Group 1 (Short) | Group 2 (Long) | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/27 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/27 | 0/28
Other Adverse Events (participants affected / at risk) | 3/28 | 1/27 | 3/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (Short) (N=28) | Group 2 (Long) (N=27) | Standard Care (N=28)
Chest pain (General disorders) | 2 (2) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 3 (3)
Motor vehicle accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes